CLINICAL TRIAL: NCT03719469
Title: Circulating microRNAs Expression as Predictors of Clinical Response in Rheumatoid Arthritis Patients Treated With Green Tea
Brief Title: Circulating microRNAs as Novel Prognosis Biomarkers for Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Sami Gabr, clinical Professor, King Saud University
Other Study IDs: RRC-2015-058
Record Dates: First submitted 2018-09-06; First posted 2018-10-25 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Rh Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — For each subject, total RNA was extracted from serum samples using the TRIzol LS reagent (Invitrogen, Carlsbad, CA), and subjected to RT-PCR analysis. A ready-made solutions containing the primers and probes for human miR-146a and miR-125ba (Applied Biosystems, Foster City, CA) and real-time RT-PCR was estimated using an ABI 7300 system (Applied Bio systems) (Mazloom et al.,2015).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Green tea group: A total of 100 subjects (aged 18-65 years) who were diagnosed as RA with moderate to severe activity at the division of rheumatology and clinical immunology at Mansoura University,After starting green tea supplement (4 to 6 cups/day; 60 to 125 mg catechins), patients were evaluated for therapeutic response at baseline and 12, and 24 weeks.
  Interventions: Dietary Supplement: Green tea group
- control group: fifty healthy normal subjects were included in this study as controls.

INTERVENTIONS:
Dietary Supplement: Green tea group
  Groups: Green tea group

SUMMARY:
The correlation of circulating serum miR-125ba and miR-146a expression and clinical response to green tea therapy were analysed in RA patients.Clinical response to green tea therapy for 24 weeks was calculated from DAS28 scores. Whereas , a decrease of 1.2 points or above in DAS28 scores at 24 weeks of treatment compared with baseline was defined as clinical response according to the EULAR response criteria.A ready-made solutions containing the primers and probes for human miR-146a and miR-125ba (Applied Biosystems, Foster City, CA) and real-time RT-PCR was estimated using an ABI 7300 system (Applied Bio systems).

DETAILED DESCRIPTION:
1. participants: A total of 100 subjects (aged 18-65 years) who were diagnosed as RA with moderate to severe activity at the division of rheumatology and clinical immunology at Mansoura University were evaluated in this study.
2. patients were evaluated for therapeutic response at baseline and 12, and 24 weeks of green tea therapy. All patients with RA were subjected for estimation of ESR, CRP, disease activity score in 28 joints (DAS28), patient's global assessment (PGA), and health assessment questionnaire damage index (HAQ-DI) at each visits (0 week, 12 weeks, and 24 weeks).
3. Pain intensity was assessed by using a standard VAS of 100 mm previously validated to chronic and acute pains.
4. Clinical response to green tea therapy for 24 weeks was calculated from DAS28 scores.
5. human miR-146a and miR-125ba were isolated and subjected to RT-PCR analysis

ELIGIBILITY:
Inclusion Criteria:

* subjects (aged 18-65 years) who were diagnosed as RA with moderate to severe activity at the division of rheumatology and clinical immunology at Mansoura University, between 20 January/2015 and 20 September 2015 were recruited in this prospective study.
* According to the diagnostic criteria of the American College of Rheumatology (Arnett et al., 1988), all patients classified as showing established RA for more than 8 years.
* Only patients who had higher scores of DAS28-ESR, RA biomarkers, and established radiographic analysis, and were diagnosed with RA according to the 2010ACR/ EULAR classification criteria were included in this study.

Exclusion Criteria:

• Patients who received non-steroidal anti-inflammatory drugs, oral glucocorticoids, had a history of severe deformation of joint, pregnant or lactating women were excluded from this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 100 subjects (aged 18-65 years) who were diagnosed as RA with moderate to severe activity at the division of rheumatology and clinical immunology at Mansoura University, between 20 January/2015 and 20 September 2015 were recruited in this prospective study. According to the diagnostic criteria of the American College of Rheumatology (Arnett et al., 1988), all patients classified as showing established RA for more than 8 years.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-01-20 (Actual); Primary Completion 2015-01-20 (Actual); Study Completion 2015-09-20 (Actual)

PRIMARY OUTCOMES:
Functional status | change from baseline functional status at 24 weeks
  It will be assessed using disease activity score -28 (DAS28) and pre-validated health assessment questionnaire damage index (HAQ-DI). For DAS28 score, the number of swelling joints count (SJC) (0-28) and tender joints count (TJC) (0-28) in all patients were examined and DAS28 scores were calculated . DAS28 values > 2.6 and ≤ 3.2 was considered as low RA disease activity, values > 3.2 and ≤ 5.1 was considered as moderate disease activity and those > 5.1 was considered as high disease activity. In case of HAQ-DI, score calculation involves answering of eight domains(dressing, rising, eating, walking, hygiene, grip, reach and usual activities) with four point likert scale . SDAI values > 3.3 and ≤11 was considered as low RA disease activity, values > 11 and ≤ 26 was considered as moderate disease activity and those > 26 was considered as high disease activity

SECONDARY OUTCOMES:
Pain intensity | change from baseline functional status at 24 weeks
  It will be assessed using the visual analogue scale (VAS). The patients were asked to mark on the VAS scale of 0-10 cm according to their global assessment of pain. The physician marked on the VAS of 0-10 cm according to the physician global assessment. Patients with higher VAS scores were considered with greater pain intensity.
Abnormal cell physiology and the parthenogenesis of Rheumatoid arthritis (RA) | change from baseline functional status at 24 weeks
  it will be assessed by estimating the role of micro ribonucleic acid (microRNAs) in maintaining immune and inflammatory responses. In this part, the expression of miRNAs was estimated by real-time polymerase chain reaction (RT-PCR) analysis, whereas serum samples of each patients were subjected to PCR analysis. Patients with higher miRNAs expressionshowed greater abnormal in cell physiology and the pathogenesis of RH. Whereas normal subjects (≤ 1.2), and abnormal subjects ( ˃ 1.2)

IPD SHARING:
Plan to Share IPD: Undecided
After starting green tea supplement (4 to 6 cups/day; 60 to 125 mg catechins), patients were evaluated for therapeutic response at baseline and 12, and 24 weeks. All patients with RA were subjected for estimation of ESR, CRP, disease activity score in 28 joints (DAS28), patient's global assessment (PGA), and health assessment questionnaire damage index (HAQ-DI) at each visits (0 week, 12 weeks, and 24 weeks). Pain intensity was assessed by using a standard VAS of 100 mm previously validated to chronic and acute pains (Aicher et al., 2012; Szyfelbein et al., 1985). Clinical response to green tea therapy for 24 weeks was calculated from DAS28 scores. Whereas , a decrease of 1.2 points or above in DAS28 scores at 24 weeks of treatment compared with baseline was defined as clinical response according to the EULAR response criteria (van Gestel et al.,1996).

REFERENCES:
- [Derived] Al-Rawaf HA, Alghadir AH, Gabr SA. MicroRNAs as Biomarkers of Pain Intensity in Patients With Chronic Fatigue Syndrome. Pain Pract. 2019 Nov;19(8):848-860. doi: 10.1111/papr.12817. Epub 2019 Aug 30. PMID 31282597